CLINICAL TRIAL: NCT01595919
Title: A Comparison of Beverages Consumed Within a Meal to Satiation on Meal-time Food Intake and Post-meal Appetite and Glycemic Response in Healthy Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, G. Harvey Anderson, Professor, University of Toronto
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: Mixed Meal Milk Study
Record Dates: First submitted 2012-05-08; First posted 2012-05-10 (Estimated); Last update posted 2012-06-15 (Estimated); Status verified 2012-06

CONDITIONS: Obesity; Hyperglycemia
MeSH Terms: conditions — Obesity; Hyperglycemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1% Milk (Experimental)
  Interventions: Other: Nutritional Intervention
- Regular Cola (Experimental)
  Interventions: Other: Nutritional Intervention
- Diet cola (Experimental)
  Interventions: Other: Nutritional Intervention
- Orange juice (Experimental)
  Interventions: Other: Nutritional Intervention
- Water (Placebo Comparator)
  Interventions: Other: Nutritional Intervention

INTERVENTIONS:
Other: Nutritional Intervention — Ad libitum amounts of beverage at a meal

SUMMARY:
The objective of the current study is to determine the effects of an ad libitum intake of 1% milk, fruit juice, regular cola, diet cola and water, as part of a pizza meal, on meal food intake, appetite and postprandial blood glucose in healthy men and women. We hypothesize that 1% milk will reduce food intake and result in better post-meal glycemic response compared to the other beverages.

ELIGIBILITY:
Inclusion Criteria:

* healthy men and women
* age 20-30 years
* BMI between 20-24.9 kg/m^2

Exclusion Criteria:

* breakfast skippers
* diabetes or any metabolic diseases
* lactose intolerance or allergies to milk
* taking medications

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2011-04; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Food Intake | 2 hours
  Measurement of energy intake during an ad libitum test meal

CONTACTS AND LOCATIONS:
Locations (1):
- University of Toronto, Department of Nutritional Sciences, Toronto, Ontario, Canada

REFERENCES:
- [Derived] El Khoury D, Panahi S, Luhovyy BL, Douglas Goff H, Harvey Anderson G. Interaction of mealtime ad libitum beverage and food intake with meal advancement in healthy young men and women. Physiol Behav. 2015 May 1;143:39-44. doi: 10.1016/j.physbeh.2015.02.023. Epub 2015 Feb 18. PMID 25700893